CLINICAL TRIAL: NCT04067024
Title: Evaluation of the Effectiveness of the Supraclavicular Block Associated With a Pecs Blocks I to Ensure Analgesia When Placing a Pacemaker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P2016/447
Record Dates: First submitted 2018-03-12; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2018-03

CONDITIONS: Pain; Pacemaker Ddd
Keywords: regional anesthesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local anesthesia by the surgeon (LAS) (Active Comparator): Local infiltration (ropivacaine 3,75 mg/ml) by surgeon
  Interventions: Procedure: Local anesthesia made by surgeon
- Regional anesthesia group (LRA): (Experimental): By ultrasound, a pecs block I associated with a supraclavicular nerf block is performed. (Ropivacaine 3,75 mg/ml)
  Interventions: Procedure: Regional anesthesia group

INTERVENTIONS:
Procedure: Local anesthesia made by surgeon — infiltration with local anesthetics
  Arms: Local anesthesia by the surgeon (LAS)
Procedure: Regional anesthesia group — Pecs block I and Supraclavicular nerf block
  Arms: Regional anesthesia group (LRA):

SUMMARY:
Pacemakers are currently placed at the Erasmus Hospital under local anesthesia performed by the surgeon, and the amount of local anesthetic agents sometimes reach the maximum permitted doses, with a risk of systemic toxicity. Moreover, these patients often present an associated conduction block. This represents a contraindication/constraint in the use of lidocaine 2% (local anesthesia frequently used by the surgeon to infiltrate). This study hypothesized that using a block of the supraclavicular nerve associated with a Pecs Block I. guided by ultrasound should require a smaller quantity of local anesthetic.

DETAILED DESCRIPTION:
PECS 1 Block and Supraclavicular Nerve Block, were performed by an anesthesiologist under ultrasound control using a linear 8Mzt transducer, a Phillips HD 11 machine and a 50 mm needle Stimuplex 360 Braun. The ALR procedure was performed 30 minutes before the surgical incision. A volume of 15 ml of ropivacaine 3.75 mg/ml is used and distributed as follows: 12 ml for the Pecs 1 Block and 3 ml for the Supraclavicular nerve block: The patient was placed in supine position with the arm abducted at about 90 °, the puncture site being sterilized with betadine. The transducer was first placed in a subclavicular position in order to identify the major and minor pectoralis muscles, as well as the thoracoacromial artery, particularly the pectoral branch, additional color Doppler, was used for the identification of those vessels. The needle was directed in plane to the intermuscular space lying between the large and small pectoral, a careful avoidance of the thoracoacromial artery or its pectoral branch was ensured. The LA injection, under visual control of the spread between the two muscles, was initiated at the level of the 2nd and 3rd ribs after a classical aspiration test; 12 ml of the ropivacaine 0.375% were used. A spread of the LA appearing as an intermuscular hypoechoic "lens" was always searched.

Second, a supraclavicular nerve block was performed. We initially identified the C5 root and scanned cranially to visualize the superficial cervical plexus. then, moving caudally, the supraclavicular nerve was isolated appearing as a hypoechogenic structure between scalenus medius and posterior border of the sternocleidomastoid muscle. A total of 3 ml of ropivacaine 0,375% was deposited nearby this nerve.

In the ALC group (Anesthesia Local Surgeon's Anesthesia: Local Infiltration of N = 15 tissues) 15 ml Ropivacaine 3.75 mg/ml were injected in the subclavicular area, as usual, starting from the skin to the depth of the muscles.

In case of patient discomfort or failure of the techniques used, a further local infiltration consisting of a maximum of 10 ml lidocaine 2% performed as required by the surgeon was allowed as rescue. If this failed, the depth of sedation would gradually increase and ventilation would be controlled either by face or laryngeal mask Propofol 1-3 mg / Kg / IV + sufentanyl 2.5 μg / IV).

ELIGIBILITY:
Inclusion Criteria:

* Women and men > 18 years of age
* Patients scheduled for the implantation of a pace-maker

Exclusion Criteria:

* Patients refusing to sign the consent
* Patients included in another protocol within 3 months
* Pregnant or breastfeeding patients
* Allergy to local anesthetics
* Patients with a contraindication to regional anesthesia (coagulopathy, local infection, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Volume of local anesthetics used | 24 hour
  ml

SECONDARY OUTCOMES:
Pain scoring | 24 hours
  Visual analog scale
Post-operative Paracetamol dose | 24h
  paracetamol mg

CONTACTS AND LOCATIONS:
Overall Officials: wendy Fernandez, Dr., Principal Investigator — Erasme Hospital,Route de lenniek 808, 1070, Brussels
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No